CLINICAL TRIAL: NCT04510701
Title: Videoscope-assisted Lateral Maxillary Sinus Floor Elevation: Evaluation of the Schneiderian Membrane for Micro-tears
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Sarah Ohnander, Principal Investigator, University of Manitoba
Other Study IDs: HS24052 (B2020:072)
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Videoscope; Maxillary Sinus; Schneiderian Membrane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: videoscope — a videoscope will be used to evaluate the integrity of the membrane while doing lateral maxillary sinus elevation surgery

SUMMARY:
This case series will recruit patients who require lateral maxillary sinus floor elevation surgery. This procedure will be carried out as per standard surgical protocol. The periodontal resident performing the surgery will evaluate the Schneiderian membrane at several points during the surgery to determine its integrity (beyond visual inspection). This will be completed by using the videoscope to evaluate the membrane. This evaluation will take place at at least 3 points during the surgery (before membrane elevation, half-way through membrane elevation, and prior to initiating bone grafting procedures). If the resident wishes to evaluate the membrane at other points during the surgery to inspect the integrity of the membrane, this may be accomplished. This evaluation will be recorded for later, further evaluation by experienced periodontists. If no visible perforation is evident, a 1% baby shampoo solution in normal saline (Johnson and Johnson) will be applied topically over the membrane prior to videoscope evaluation. At this point, the patient will lightly blow their nose; if any micro-tears not visible to the naked eye are present, these tears will produce a bubbling effect, which will be recorded by the videoscope. This evaluation will take place with the 1st and 2nd videoscope evaluations (before membrane elevation, and mid-way through elevation).

Patients will be asked to complete a VAS questionnaire at their one-week follow-up appointment in order to determine how post-op healing has been progressing.

After all procedures have been performed, three experienced periodontists will individually evaluate the videos post-surgically. They will evaluate each video and determine if, in their opinion, there is a membrane perforation (yes/no). Each video will be evaluated in a random fashion (each video being evaluated as a separate event, and not by case). The evaluating periodontists will also be masked to the results noted by the surgeon who completed the surgery, and blinded to the patient's information.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring maxillary sinus floor elevation (lateral approach), with current subantral bone height 6 mm or less
* Male or female patient, 18 years of age and older
* Patients who exhibit adequate ability to comply with postoperative instructions, research protocols and methods
* Patients who have read, understand, and have signed the informed consent form
* Patients with an adequate level of oral hygiene, defined as Full Mouth Plaque Score (FMPS) and Full Mouth Bleeding Score (FMBS) should be <20% (after periodontal therapy, if necessary)

Exclusion Criteria:

Absolute contraindications:

* Patients on IV bisphosphonates
* Patients who are undergoing chemotherapy
* Patients who have undergone head and neck radiotherapy where the field of irradiation included the maxilla
* Patients whose membrane thickness is increased due to an existing sinus pathology (sinusitis or mucosal cysts): These conditions should be treated prior to surgical treatment (S. W. Kim et al. 2019)
* Diabetic patients with uncontrolled diabetes and poor glycemic control
* Patients who are undergoing long-term immunosuppressive therapy, or have been taking corticosteroids long-term (Bornstein et al. 2009)
* Patients with active or untreated periodontitis

Relative contraindications:

* Patients who have been receiving long term oral bisphosphonate therapy (3 years duration or more) (Bornstein et al. 2009)
* Patients who smoke >10 cigarettes per day
* Patients who are alcohol abusers (Li and Wang 2008)
* Patients who are on antithrombotic medications should be treated with extra caution during surgery, as well as patients with blood disorders that may affect hemostasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Dr. Sam Borden Graduate Periodontics Clinic, Dr. Gerald Niznick College of Dentistry, University of Manitoba who require lateral sinus floor elevation surgery.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
incidence of micro-tears present in the Schneiderian membrane | first evaluation will be done before the membrane is elevated; second will be part-way through elevation of the membrane; and the third evaluation will be once membrane elevation has been completed
  incidence of micro-tears will be evaluated at 3 points during the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada